CLINICAL TRIAL: NCT05775003
Title: Effects of Adding L-BAIBA or L-BAIBA + Grains of Paradise to Exercising Adult Overweight and Obese Men and Women on Changes in Body Composition, Resting Metabolic, and Cardiometabolic Risk Factors
Brief Title: Effects of Adding L-BAIBA or L-BAIBA + Grains of Paradise to Exercising Adult Overweight and Obese Men and Women
Acronym: GOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-23-28
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obese; Weight Loss; Body Weight; Cardiometabolic Syndrome
Keywords: weight loss; body composition; cardiometabolic syndrome
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will be conducted using a double-blind, placebo-controlled, parallel group design. Eligible study participants will be randomly assigned to one of three supplementation groups: placebo (resistant starch) supplementation + exercise group, 500 mg BAIBA supplementation + exercise group, and a 500 mg BAIBA supplementation + 40 mg Grains of Paradise + exercise group.
Who Masked: Participant, Investigator
Masking Description: Eligible study participants will be randomly assigned to one of three supplementation groups: placebo (resistant starch) supplementation + exercise group, 500 mg BAIBA supplementation + exercise group, and a 500 mg BAIBA supplementation + 40 mg Grains of Paradise + exercise group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Resistant starch
  Interventions: Dietary Supplement: Exercise
- 500 mg BAIBA supplementation (Experimental): 500 mg BAIBA supplementation
  Interventions: Dietary Supplement: Exercise
- 500 mg BAIBA supplementation + 40 mg Grains of Paradise (Experimental): 500 mg BAIBA supplementation + 40 mg Grains of Paradise
  Interventions: Dietary Supplement: Exercise

INTERVENTIONS:
Dietary Supplement: Exercise — 8 week exercise training program - consisting of weight training and cardiovascular exercise
  Other Names: Exercise training

SUMMARY:
The goal of this intervention study is to examine changes in body composition, weight loss, and cardio-metabolic risk factors after adding supplementation of L-Beta aminoisobutyric acid (L-BAIBA) and Grains of Paradise to exercise in overweight and obese men and women. Participants will supplement for 8 weeks and complete a 8 week exercise protocol.

DETAILED DESCRIPTION:
This study will be conducted using a double-blind, placebo-controlled, parallel group design. Eligible study participants will be randomly assigned to one of three supplementation groups: placebo (resistant starch) supplementation + exercise group, 500 mg BAIBA supplementation + exercise group, and a 500 mg BAIBA supplementation + 40 mg Grains of Paradise + exercise group. After signing an IRB-approved consent form, prospective participants will be scheduled for a screening visit where they will have their eligibility finalized through completion of a peak VO2 assessment using a motorized treadmill and metabolic cart. Eligible participants will then be fully explained the study and scheduled for a baseline testing session (week 0). Prior to scheduling this visit, participants must complete a 4-day food record. Once a food record is completed, participants will observe an overnight fast and be scheduled to complete the testing session between the hours of 0600 - 1000 hours. Upon arrival, changes in medical status, medications, and dietary supplements will be confirmed before having their body mass and hemodynamics assessed. After hemodynamic assessment, participants will have the first of two resting metabolic rate measurements completed before having a venous blood sample collected for evaluation of health markers (complete blood counts, comprehensive metabolic panels, and lipid panels). Participants will then use an electronic tablet and complete the Profile of Mood States and visual analog scales to evaluate perceptions of energy, focus, attention, hunger, appetite, and concentration. Participants will then be given their daily dose and a timer will be started. From there, participants will have their waist circumference, body water (BIS), and body composition (DEXA) assessed. After completion of these, participants will then wait in the laboratory until an hour has passed and will have a second resting metabolic rate measurement completed. After the second resting metabolic rate measurement, participants will have a second venous blood sample collected to evaluate changes in glycerol. All participants will be given instructions and meal plans as well as be offered weekly educational sessions on how to restrict calories and meet protein goals throughout the study protocol. Participants will complete five days per week of exercise consisting of a mixture of walking and resistance training. Daily compliance to the exercise and supplementation groups will be monitored weekly for an 8-week period. Participants who complete at least 80% of their assigned workouts will be considered compliant and will be scheduled for follow-up visits after 2, 4, and 8 weeks of supplementation.

Participants will be asked to follow an 8-10 hour dry fast and to refrain from caffeine, alcohol, nicotine, and exercise (excluding the 30 min daily walk) for 24 hours prior to each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are between 18 - 60 years of age
* Body mass index values will range from >25.0 to < 32.0 kg/m2, making them qualified as an overweight-to-obese population (https://www.nhlbi.nih.gov/health/educational/lose_wt/BMI/bmicalc.htm)
* Average body mass index for entire study cohort will be less than 30.0 kg/m2. As such an ongoing calculation of the recruited cohort's mean body mass index will be maintained and people will only be randomized into the study if the average cohort body mass index value does not exceed 30.0 kg/m2
* Free-living/uninhibited with use of ambulatory assistive devices (e.g. canes, crutches, walkers, etc.) and independent
* In good health absent of being overweight or mildly obese with no other signs or symptoms of cardiovascular, respiratory, metabolic, immune, psychiatric, or musculoskeletal disease or disorders
* Willingness to maintain consistent sleep duration the evening before study visits
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, and carry out all study-related procedures
* Able to complete a peak oxygen consumption exercise test with no contraindications to perform exercise per standards put forth by the American
* College of Sports Medicine. In other words, they are able to safety complete maximal exercise.

Exclusion Criteria:

* Positive medical history and/or is currently being treated for some form of heart disease, cardiovascular disease
* Currently being treated for kidney disease, renal failure, or has dialysis performed on regular intervals
* Has liver disease or some form of clinically diagnosed hepatic impairment
* Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL)
* Diagnosed with or is being treated for some form of thyroid disease
* Diagnosed with major affective disorder or other psychiatric disorder that required hospitalization in the prior year
* Diagnosed with some form of immune disorder (i.e., HIV/AIDS)
* History of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
* Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
* Positive medical history for any neurological condition or neurological disease
* Currently prescribed a statin drugs (i.e., Lipitor, Livalo, Crestor, Zocor, etc.) or any hypertension medications (i.e., Beta-blockers, ACE Inhibitors, Alpha blockers, Vasodilators, etc.)
* Current smoker (average of > 1 pack per day within the past 3 months) or has quit within the past six months. This includes all forms of nicotine
* Intake of any drugs (prescribed or over the counter) or dietary supplements that are known or are purported to weight loss such as thermogenics, hydroxycitric acid, ephedra, capsaicin, etc.
* Participants who are lactating, pregnant or planning to become pregnant
* Have a known sensitivity or allergy to any of the study products
* History of alcohol or substance abuse in the 12 months prior to screening
* Receipt or use of an investigational product in another research study within 30 days of beginning the study protocol
* They plan major changes in lifestyle (i.e., diet, dieting, exercise level, travel, etc.) during the study
* Recent history (<3 months) of exercise training or weight loss (> 5%)
* Any orthopedic limitation that would prevent participation in a general fitness program
* Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Fat Mass (4-Compartment) | 8 Weeks
  Changes in fat mass using a 4 compartment model

SECONDARY OUTCOMES:
Lean mass (4-Compartment) | 8 weeks
  changes in lean mass using a 4 compartment model
Waist circumference | 8 weeks
  Changes in waist circumference
Visceral Fat (DEXA) | 8 weeks
  Changes in Visceral Fat (DEXA)
Lean:Fat Ratio (DEXA) | 8 weeks
  Changes in Lean:Fat Ratio (DEXA)
Body Mass | 8 weeks
  Changes in Body Mass
Hunger and appetite visual analog scale | 8 weeks
  Changes in Hunger and appetite visual analog scale. Minimum score is 0. Maximum score is 100. Lower is better.
Energy, focus, attention, and concentration visual analog scales | 8 weeks
  Changes in Energy, focus, attention, and concentration visual analog scales. Minimum score is 0. Maximum score is 100. Higher is better.
Profile of mood states (POMS) | 8 weeks
  Changes in Profile of mood states (POMS) Minimum score is 0. Maximum score is 5 for each question. A higher Total Mood Disturbance score is worse, lower is better.
Serum Glycerol | 8 weeks
  Changes in Serum Glycerol Levels
Fasting glucose | 8 weeks
  Changes in Fasting glucose
Complete Blood Count | 8 weeks
  Changes in Complete Blood Count
Comprehensive Metabolic Panel | 8 weeks
  Changes in Comprehensive Metabolic Panel
Lipid Panel | 8 weeks
  Changes in Lipid Panel
Self-reported adverse events | 8 weeks
  Occurrences of Self-reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Layman DK, Evans E, Baum JI, Seyler J, Erickson DJ, Boileau RA. Dietary protein and exercise have additive effects on body composition during weight loss in adult women. J Nutr. 2005 Aug;135(8):1903-10. doi: 10.1093/jn/135.8.1903. PMID 16046715
- [Background] Kerksick C, Thomas A, Campbell B, Taylor L, Wilborn C, Marcello B, Roberts M, Pfau E, Grimstvedt M, Opusunju J, Magrans-Courtney T, Rasmussen C, Wilson R, Kreider RB. Effects of a popular exercise and weight loss program on weight loss, body composition, energy expenditure and health in obese women. Nutr Metab (Lond). 2009 May 14;6:23. doi: 10.1186/1743-7075-6-23. PMID 19442301
- [Background] Kerksick CM, Wismann-Bunn J, Fogt D, Thomas AR, Taylor L, Campbell BI, Wilborn CD, Harvey T, Roberts MD, La Bounty P, Galbreath M, Marcello B, Rasmussen CJ, Kreider RB. Changes in weight loss, body composition and cardiovascular disease risk after altering macronutrient distributions during a regular exercise program in obese women. Nutr J. 2010 Nov 22;9:59. doi: 10.1186/1475-2891-9-59. PMID 21092228
- [Background] Kerksick CM, Roberts MD, Campbell BI, Galbreath MM, Taylor LW, Wilborn CD, Lee A, Dove J, Bunn JW, Rasmussen CJ, Kreider RB. Differential Impact of Calcium and Vitamin D on Body Composition Changes in Post-Menopausal Women Following a Restricted Energy Diet and Exercise Program. Nutrients. 2020 Mar 7;12(3):713. doi: 10.3390/nu12030713. PMID 32156010
- [Background] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845
- [Background] Wilson JP, Fan B, Shepherd JA. Total and regional body volumes derived from dual-energy X-ray absorptiometry output. J Clin Densitom. 2013 Jul-Sep;16(3):368-373. doi: 10.1016/j.jocd.2012.11.001. Epub 2013 Jan 12. PMID 23321490
- [Background] Smith-Ryan AE, Mock MG, Ryan ED, Gerstner GR, Trexler ET, Hirsch KR. Validity and reliability of a 4-compartment body composition model using dual energy x-ray absorptiometry-derived body volume. Clin Nutr. 2017 Jun;36(3):825-830. doi: 10.1016/j.clnu.2016.05.006. Epub 2016 May 15. PMID 27237796